CLINICAL TRIAL: NCT02312687
Title: A Phase 2b, Open-Label, Long-Term Extension Study to Evaluate the Safety and Pharmacodynamics of KRN23 in Adult Subjects With X-Linked Hypophosphatemia (XLH)
Brief Title: Long-Term Extension Study of KRN23 in Adult Subjects With X-Linked Hypophosphatemia (XLH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX023-CL203
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2014-12-03; First posted 2014-12-09 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: X-Linked Hypophosphatemia
Keywords: XLH; FGF23; KRN23
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KRN23 (Experimental): KRN23 subcutaneous (SC) injections every 4 weeks. Starting doses will be based on the subject's last dose in study KRN23-INT-001 (NCT02312687) or KRN23-INT-002 (NCT01571596). Doses may be titrated to achieve the target peak serum phosphorus range.
  Interventions: Biological: KRN23

INTERVENTIONS:
Biological: KRN23 — solution for SC injection
  Other Names: burosumab; Crysvita®

SUMMARY:
The primary objectives of this study are to:

* Assess the long-term safety of KRN23 subcutaneous (SC) administration in adult subjects with XLH
* Assess the proportion of subjects achieving serum phosphorus levels in the normal range (2.5-4.5 mg/dL) with long-term administration of KRN23
* Assess long-term pharmacodynamics (PD) of KRN23 as measured by changes in the following: serum intact parathyroid hormone (iPTH); serum and urinary phosphorus; ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate (TmP/GFR) and tubular reabsorption of phosphate (TRP); serum 1,25-dihydroxy vitamin D (1,25[OH]2D); serum fibroblast growth factor 23 (FGF23); bone biomarkers: serum alkaline phosphatase (ALP), bone-specific ALP (BALP), carboxy terminal crosslinked telopeptide of type I collagen (CTx), and procollagen type 1 N-terminal propeptide (P1NP)
* Assess long-term immunogenicity of KRN23 as measured by presence of anti-KRN23 antibody (ADA)

ELIGIBILITY:
Inclusion Criteria:

1. Have participated in Kyowa Hakko Kirin Pharma, Inc.'s KRN23-INT-001 (NCT01340482) or KRN23-INT-002 (NCT01571596) studies (received at least 2 doses of KRN23)
2. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min or eGFR of 45 to < 60 mL/min at Screening with confirmation that the renal insufficiency was not due to nephrocalcinosis.
3. Sexually active subjects must be willing to use an acceptable method of contraception (e.g., double barrier method) while participating in the study and for 30 days after receiving the last dose of KRN23.

Exclusion Criteria:

1. Subject experienced a safety-related event in the KRN23-INT-001 or KRN23-INT-002 study that, in the opinion of the investigator and sponsor, precludes resuming KRN23 treatment.
2. Presence of nephrocalcinosis on renal ultrasound that, in the opinion of the investigator and sponsor, precludes resuming KRN23 treatment.
3. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
4. Participation in an investigational drug or device trial within 30 days of enrollment (other than KRN23-INT-001 or KRN23-INT-002).
5. Use of a pharmacologic vitamin D metabolite or analog (e.g., calcitriol, doxercalciferol, and paricalcitol), phosphate, or aluminum hydroxide antacids (e.g., Maalox® and Mylanta®) within 21 days prior to Screening or during the study.
6. Use of medication to suppress parathyroid hormone (PTH) (e.g., Sensipar®, cinacalcet, calcimimetics) within 2 months prior to Screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- United States (5):
  - University California San Francisco Hospital, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University Hospital, Indianapolis, Indiana
  - Duke University, Durham, North Carolina
  - Houston Methodist Reasearch Institute, Houston, Texas

REFERENCES:
- [Derived] Weber TJ, Imel EA, Carpenter TO, Peacock M, Portale AA, Hetzer J, Merritt JL, Insogna K. Long-term Burosumab Administration Is Safe and Effective in Adults With X-linked Hypophosphatemia. J Clin Endocrinol Metab. 2022 Dec 17;108(1):155-165. doi: 10.1210/clinem/dgac518. PMID 36072994

RESULTS

PARTICIPANT FLOW:
Groups:
- KRN23: KRN23 subcutaneous (SC) injections every 4 weeks
Period: Overall Study
Arm/Group | KRN23
Started | 20
Completed | 19
Not Completed | 1
Not completed — Other, Not Specified | 1

BASELINE CHARACTERISTICS:
Groups:
- KRN23: KRN23 SC injections every 4 weeks
Arm/Group | KRN23
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 1.89 (0.301)
Serum Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pg/mL] | 110.8 (43.70)
Serum Total Fibroblast Growth Factor 23 (FGF23) [Mean (Standard Deviation); unit: pg/mL] | 262.9 (227.02)
Serum Free FGF23 [Mean (Standard Deviation); unit: pg/mL] | 81.9 (42.33)
Serum 1,25-dihydroxy vitamin D [1,25(OH)2D] [Mean (Standard Deviation); unit: pg/mL] | 31.7 (12.61)
2-hour Urine TmP/GFR [Mean (Standard Deviation); unit: mg/dL] — TmP/GFR: ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate
  mg/dL | 1.583 (0.2566)
2-hour Urine Tubular Reabsorption of Phosphate (TRP) [Mean (Standard Deviation); unit: fraction of phosphorus reabsorbed] | 0.783 (0.0792)
Fractional Excretion of Phosphorus (FEP) [Mean (Standard Deviation); unit: fraction of phosphorus excreted] | 0.217 (0.0792)
24-hour Urine Phosphorus [Mean (Standard Deviation); unit: g/24hr] | 0.74 (0.322)
24-Hour Urine Calcium [Mean (Standard Deviation); unit: mg/24hr] — Population: participants with an assessment
  mg/24hr
    number analyzed (Participants) | 17
    (all) | 96.118 (75.9530)
24-Hour Urine Creatinine [Mean (Standard Deviation); unit: mg/24hr] | 1058.150 (444.3073)
24-Hour Urine Calcium/Creatinine Ratio [Mean (Standard Deviation); unit: mg/mg] — Population: participants with an assessment
  mg/mg
    number analyzed (Participants) | 17
    (all) | 0.0881 (0.05034)
Total Alkaline Phosphatase (ALP) [Mean (Standard Deviation); unit: U/L] | 131.1 (50.50)
Bone-Specific Alkaline Phosphatase (BALP) [Mean (Standard Deviation); unit: mcg/L] | 31.26 (18.528)
Carboxy Terminal Cross-Linked Telopeptide of Type I Collagen (CTx) [Mean (Standard Deviation); unit: pg/mL] | 732.4 (404.01)
Procollagen Type N-Propeptide (P1NP) [Mean (Standard Deviation); unit: ng/mL] | 76.5 (41.58)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Treatment Emergent AEs (TEAEs), Serious AEs (SAEs), and AEs Leading to Discontinuation or Death
Description: An AE is defined as any untoward medical occurrence, whether or not considered drug related. An SAE or serious suspected adverse reaction is an AE or suspected adverse reaction that at any dose, in the view of either the investigator or sponsor, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect; an important medical event. A TEAE is an AE that occurred on or after the first burosumab dose. AEs were graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). AEs were classified by the Investigator as possibly related, probably related, or definitely related.
Time Frame: Screening through the end of study plus 4-8 weeks. The mean duration of burosumab exposure was 165.6 weeks (range: 68-184 weeks).
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  All AEs | 20
  TEAEs | 20
  Related AEs | 12
  SAEs | 9
  Related SAEs | 1
  Grade 3 and 4 AEs | 10
  AEs Leading to Discontinuation | 0
  AEs Leading to Death | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  Hypertension | 2
  Decreased blood pressure | 1

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Values, by Category
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  Elevated eosinophils | 1
  Hypercholesterolemia | 1
  Hyperkalemia | 1
  Hyperglycemia | 1
  Elevated alanine aminotransferase | 1
  Elevated aspartate aminotransferase | 1
  Elevated gamma-glutamyl transferase | 2
  Proteinuria | 2
  Elevated amylase | 2
  Elevated alkaline phosphatase | 1
  Elevated lipase | 1
  Hypercalciuria | 1
  Worsening hypercholesterolemia | 2
  Decreased hemoglobin | 2
  Hypocalcemia (intermittent) | 1
  Hypovitaminosis D | 1
  Elevated cholesterol | 1
  Hyperparathyroidism | 1
  Urine electrophoresis abnormal | 1

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Exams, by Category
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  Bone pain | 1
  Conjunctival haemorrhage | 1
  Hypoacusis | 1
  Dermal cyst | 1
  Osteoarthritis | 1
  Gravitational oedema | 1
  Hypoaesthesia | 1
  Neuropathy peripheral | 2
  Arthralgia | 1
  Peroneal nerve palsy | 1
  Spinal pain | 1
  Bone lesion | 1
  Femur fracture | 1
  Scrotal oedema | 1
  Synovial cyst | 1
  Testicular swelling | 1
  Thermal burn | 1
  Weight decreased | 1

5. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Echocardiogram (ECHO) Tests
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in ECGs
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Renal Ultrasound, by Category
Description: Clinically significant changes from baseline reported as adverse events are presented.
Time Frame: Through Week 184
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  Kidney stone(s) | 1
  Nephrocalcinosis | 1
  Right renal mass | 1
  Nephrolithiasis | 2

8. Primary Outcome: Number of Participants Positive for Anti-KRN23 Antibodies and Neutralizing Antibodies at Baseline and Anytime Post-Baseline
Time Frame: Through Week 184
Population: Participants tested for neutralizing antibodies (n=4) are those who were positive for anti-KRN23 antibodies at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
Participants
  Baseline: Anti-KRN23 Antibodies | 2
  Post Baseline:Anti-KRN23 Antibodies | 4
  Baseline: Neutralizing Antibodies: number analyzed (Participants) | 2
  Baseline: Neutralizing Antibodies | 0
  Postbaseline: Neutralizing Antibodies: number analyzed (Participants) | 4
  Postbaseline: Neutralizing Antibodies | 0

9. Primary Outcome: Percentage of Participants Reaching Serum Phosphorus Normal Range at Baseline and Any Time After Dosing
Time Frame: Through Week 184
Population: Pharmacodynamic (PD) Analysis Set: all participants who received at least 1 dose of burosumab and had evaluable serum/urinary data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KRN23
Number analyzed (Participants) | 20
percentage of participants | 100 [83.9 to 100.0]

10. Primary Outcome: Change From Baseline Over Time in Serum Phosphorus
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: PD Analysis Set (all participants who received at least 1 dose of burosumab and had evaluable serum/urinary data) with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | KRN23
Number analyzed (Participants) | 20
mg/dL
  Change at Week 24: number analyzed (Participants) | 16
  Change at Week 24 | 0.68 (0.103)
  Change at Week 48: number analyzed (Participants) | 19
  Change at Week 48 | 0.68 (0.055)
  Change at Week 72 | 0.59 (0.077)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 0.47 (0.081)
  Change at Week 120: number analyzed (Participants) | 18
  Change at Week 120 | 0.57 (0.082)
  Change at Week 144: number analyzed (Participants) | 18
  Change at Week 144 | 0.59 (0.084)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p < 0.0001, generalized estimation equation (GEE) — The generalized estimation equation (GEE) model includes the change from baseline as the dependent variable, time as the categorical variable and adjusted for baseline measurement, with compound symmetry covariance structure; Least Squares (LS) Mean = 0.68, 95% CI 2-sided [0.48 to 0.88]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p < 0.0001, GEE — The GEE model includes the change from baseline as the dependent variable, time as the categorical variable and adjusted for baseline measurement, with compound symmetry covariance structure; LS Mean = 0.68, 95% CI 2-sided [0.57 to 0.79]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 0.59, 95% CI 2-sided [0.44 to 0.75]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 0.47, 95% CI 2-sided [0.31 to 0.63]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 0.57, 95% CI 2-sided [0.41 to 0.73]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 0.59, 95% CI 2-sided [0.43 to 0.76]

11. Primary Outcome: Change From Baseline Over Time in Serum iPTH
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
pg/mL
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | -9.75 (6.551)
  Change at Week 48 | -11.17 (7.444)
  Change at Week 72 | -18.12 (4.567)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -25.28 (5.577)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -22.39 (4.655)
  Change at Week 144: number analyzed (Participants) | 19
  Change at Week 144 | -28.33 (6.007)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p = 0.1366, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -9.75, 95% CI 2-sided [-22.59 to 3.09]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p = 0.1334, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -11.17, 95% CI 2-sided [-25.76 to 3.42]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -18.12, 95% CI 2-sided [-27.07 to -9.17]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -25.28, 95% CI 2-sided [-36.21 to -14.35]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p < 0.0001, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -22.39, 95% CI 2-sided [-31.51 to -13.26]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE estimate — [p-value comment as in outcome 10, analysis 2]; LS Mean = -28.33, 95% CI 2-sided [-40.11 to -16.56]

12. Primary Outcome: Change From Baseline Over Time in Serum Total FGF23
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
pg/mL
  Change at Week 24 | 215493.38 (10634.172)
  Change at Week 48 | 202525.38 (17429.124)
  Change at Week 72 | 221481.03 (21353.941)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 221674.07 (20592.592)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | 208270.02 (20945.303)
  Change at Week 144: number analyzed (Participants) | 17
  Change at Week 144 | 235953.55 (35634.821)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 215493.38, 95% CI 2-sided [194650.78 to 236335.97]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 202525.38, 95% CI 2-sided [168364.92 to 236685.83]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 221481.03, 95% CI 2-sided [179628.07 to 263333.98]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 221674.07, 95% CI 2-sided [181313.34 to 262034.81]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 208270.02, 95% CI 2-sided [167217.98 to 249322.06]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 235953.55, 95% CI 2-sided [166110.59 to 305796.52]

13. Primary Outcome: Change From Baseline Over Time in Serum Free FGF23
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
pg/mL
  Change at Week 24 | 1277.84 (38.521)
  Change at Week 48 | 1244.99 (40.250)
  Change at Week 72 | 1298.49 (33.129)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 1311.05 (37.119)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | 1368.68 (21.063)
  Change at Week 144: number analyzed (Participants) | 17
  Change at Week 144 | 1298.41 (45.972)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1277.84, 95% CI 2-sided [1202.34 to 1353.34]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1244.99, 95% CI 2-sided [1166.10 to 1323.88]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1298.49, 95% CI 2-sided [1233.56 to 1363.43]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1311.05, 95% CI 2-sided [1238.30 to 1383.80]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1368.68, 95% CI 2-sided [1327.40 to 1409.96]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 1298.41, 95% CI 2-sided [1208.31 to 1388.51]

14. Primary Outcome: Change From Baseline Over Time in Serum 1,25(OH)2D
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
pg/mL
  Change at Week 24 | 7.87 (2.403)
  Change at Week 48: number analyzed (Participants) | 19
  Change at Week 48 | 2.70 (2.653)
  Change at Week 72 | 2.62 (2.505)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 0.31 (2.052)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -0.48 (2.365)
  Change at Week 144: number analyzed (Participants) | 19
  Change at Week 144 | -3.43 (2.844)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p = 0.0011, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 7.87, 95% CI 2-sided [3.16 to 12.58]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p = 0.3092, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 2.70, 95% CI 2-sided [-2.50 to 7.90]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p = 0.2958, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 2.62, 95% CI 2-sided [-2.29 to 7.53]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p = 0.8796, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 0.31, 95% CI 2-sided [-3.71 to 4.33]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p = 0.8396, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -0.48, 95% CI 2-sided [-5.11 to 4.16]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p = 0.2284, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -3.43, 95% CI 2-sided [-9.00 to 2.15]

15. Primary Outcome: Change From Baseline Ovr Time in 2-hour Urine TmP/GFR
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | KRN23
Number analyzed (Participants) | 20
mg/dL
  Change at Week 24: number analyzed (Participants) | 16
  Change at Week 24 | 0.57 (0.128)
  Change at Week 48: number analyzed (Participants) | 19
  Change at Week 48 | 0.47 (0.047)
  Change at Week 72 | 0.42 (0.072)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 0.44 (0.084)
  Change at Week 120: number analyzed (Participants) | 18
  Change at Week 120 | 0.36 (0.066)
  Change at Week 144: number analyzed (Participants) | 18
  Change at Week 144 | 0.47 (0.078)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = 0.57, 95% CI 2-sided [0.32 to 0.83]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = 0.47, 95% CI 2-sided [0.37 to 0.56]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = 0.42, 95% CI 2-sided [0.28 to 0.56]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = 0.44, 95% CI 2-sided [0.27 to 0.60]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = 0.36, 95% CI 2-sided [0.23 to 0.48]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = 0.47, 95% CI 2-sided [0.32 to 0.62]

16. Primary Outcome: Change From Baseline Over Time in in 2-hour Urine TRP
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: fraction of phosphorus reabsorbed
Arm/Group | KRN23
Number analyzed (Participants) | 20
fraction of phosphorus reabsorbed
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | 0.04 (0.015)
  Change at Week 48: number analyzed (Participants) | 19
  Change at Week 48 | 0.01 (0.011)
  Change at Week 72 | 0.01 (0.011)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 0.05 (0.012)
  Change at Week 120: number analyzed (Participants) | 18
  Change at Week 120 | 0.01 (0.012)
  Change at Week 144: number analyzed (Participants) | 18
  Change at Week 144 | 0.02 (0.017)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = 0.04, 95% CI 2-sided [0.01 to 0.07]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = 0.01, 95% CI 2-sided [-0.01 to 0.04]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = 0.05, 95% CI 2-sided [0.02 to 0.07]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = 0.01, 95% CI 2-sided [-0.02 to 0.03]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = 0.02, 95% CI 2-sided [-0.01 to 0.05]

17. Primary Outcome: Change From Baseline Over Time in FEP
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: fraction of phosphorus excreted
Arm/Group | KRN23
Number analyzed (Participants) | 20
fraction of phosphorus excreted
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | -0.04 (0.015)
  Change at Week 48: number analyzed (Participants) | 19
  Change at Week 48 | -0.01 (0.011)
  Change at Week 72 | -0.01 (0.011)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -0.05 (0.012)
  Change at Week 120: number analyzed (Participants) | 18
  Change at Week 120 | -0.01 (0.012)
  Change at Week 144: number analyzed (Participants) | 18
  Change at Week 144 | -0.02 (0.017)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = -0.04, 95% CI 2-sided [-0.07 to -0.01]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.03 to 0.01]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.04 to 0.01]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = -0.05, 95% CI 2-sided [-0.07 to -0.02]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.03 to 0.02]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = -0.02, 95% CI 2-sided [-0.05 to 0.01]

18. Primary Outcome: Change From Baseline Over Time in 24-hour Urine Phosphorus
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: g/24hr
Arm/Group | KRN23
Number analyzed (Participants) | 20
g/24hr
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | -0.01 (0.045)
  Change at Week 48 | 0.02 (0.044)
  Change at Week 72: number analyzed (Participants) | 19
  Change at Week 72 | 0.08 (0.044)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -0.01 (0.040)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -0.01 (0.058)
  Change at Week 144: number analyzed (Participants) | 16
  Change at Week 144 | -0.05 (0.054)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.10 to 0.08]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = 0.02, 95% CI 2-sided [-0.07 to 0.10]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = 0.08, 95% CI 2-sided [-0.01 to 0.16]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.09 to 0.06]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.12 to 0.10]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = -0.05, 95% CI 2-sided [-0.16 to 0.06]

19. Primary Outcome: Change From Baseline Over Time in 24-Hour Urine Calcium
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mg/24hr
Arm/Group | KRN23
Number analyzed (Participants) | 20
mg/24hr
  Change at Week 24: number analyzed (Participants) | 13
  Change at Week 24 | 22.89 (12.605)
  Change at Week 48: number analyzed (Participants) | 15
  Change at Week 48 | 15.15 (8.914)
  Change at Week 72: number analyzed (Participants) | 14
  Change at Week 72 | 11.10 (12.975)
  Change at Week 96: number analyzed (Participants) | 12
  Change at Week 96 | -16.65 (10.637)
  Change at Week 120: number analyzed (Participants) | 13
  Change at Week 120 | 3.48 (18.375)
  Change at Week 144: number analyzed (Participants) | 14
  Change at Week 144 | 28.55 (20.239)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = 22.89, 95% CI 2-sided [-1.81 to 47.60]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = 15.15, 95% CI 2-sided [-2.32 to 32.62]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = 11.10, 95% CI 2-sided [-14.33 to 36.53]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = -16.65, 95% CI 2-sided [-37.50 to 4.20]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = 3.48, 95% CI 2-sided [-32.53 to 39.49]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = 28.55, 95% CI 2-sided [-11.12 to 68.22]

20. Primary Outcome: Change From Baseline Over Time in 24-Hour Urine Creatinine
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mg/24hr
Arm/Group | KRN23
Number analyzed (Participants) | 20
mg/24hr
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | -14.77 (37.170)
  Change at Week 48 | -70.79 (46.186)
  Change at Week 72: number analyzed (Participants) | 19
  Change at Week 72 | -16.11 (48.389)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -41.74 (55.546)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -76.11 (82.239)
  Change at Week 144: number analyzed (Participants) | 17
  Change at Week 144 | -96.06 (56.389)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = -14.77, 95% CI 2-sided [-87.62 to 58.08]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = -70.79, 95% CI 2-sided [-161.31 to 19.74]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = -16.11, 95% CI 2-sided [-110.96 to 78.73]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = -41.74, 95% CI 2-sided [-150.61 to 67.13]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = -76.11, 95% CI 2-sided [-237.29 to 85.08]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = -96.06, 95% CI 2-sided [-206.59 to 14.46]

21. Primary Outcome: Change From Baseline Over Time in 24-Hour Urine Calcium/Creatinine Ratio
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mg/mg
Arm/Group | KRN23
Number analyzed (Participants) | 20
mg/mg
  Change at Week 24: number analyzed (Participants) | 13
  Change at Week 24 | 0.01 (0.010)
  Change at Week 48: number analyzed (Participants) | 15
  Change at Week 48 | 0.01 (0.011)
  Change at Week 72: number analyzed (Participants) | 14
  Change at Week 72 | 0.00 (0.011)
  Change at Week 96: number analyzed (Participants) | 12
  Change at Week 96 | -0.01 (0.013)
  Change at Week 120: number analyzed (Participants) | 13
  Change at Week 120 | 0.00 (0.013)
  Change at Week 144: number analyzed (Participants) | 14
  Change at Week 144 | 0.03 (0.023)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; LS Mean = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; LS Mean = 0.01, 95% CI 2-sided [-0.01 to 0.04]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; LS Mean = 0.00, 95% CI 2-sided [-0.02 to 0.02]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; LS Mean = -0.01, 95% CI 2-sided [-0.04 to 0.02]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; LS Mean = 0.00, 95% CI 2-sided [-0.02 to 0.03]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; LS Mean = 0.03, 95% CI 2-sided [-0.01 to 0.08]

22. Primary Outcome: Change From Baseline Over Time in Total ALP
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | KRN23
Number analyzed (Participants) | 20
U/L
  Change at Week 24 | 14.92 (6.935)
  Change at Week 48 | -1.73 (5.752)
  Change at Week 72 | -22.28 (4.044)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -20.93 (3.567)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -18.77 (7.228)
  Change at Week 144: number analyzed (Participants) | 19
  Change at Week 144 | -25.72 (5.701)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p = 0.0314, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 14.92, 95% CI 2-sided [1.33 to 28.52]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p = 0.7640, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -1.73, 95% CI 2-sided [-13.00 to 9.55]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -22.28, 95% CI 2-sided [-30.20 to -14.35]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -20.93, 95% CI 2-sided [-27.92 to -13.94]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p = 0.0094, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -18.77, 95% CI 2-sided [-32.93 to -4.60]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -25.72, 95% CI 2-sided [-36.89 to -14.54]

23. Primary Outcome: Change From Baseline Over Time in BALP
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mcg/L
Arm/Group | KRN23
Number analyzed (Participants) | 20
mcg/L
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | 4.68 (3.389)
  Change at Week 48 | -2.68 (2.247)
  Change at Week 72: number analyzed (Participants) | 19
  Change at Week 72 | -7.45 (1.067)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -8.08 (0.910)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -10.01 (1.561)
  Change at Week 144: number analyzed (Participants) | 16
  Change at Week 144 | -10.89 (1.979)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p = 0.1673, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 4.68, 95% CI 2-sided [-1.96 to 11.32]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p = 0.2330, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -2.68, 95% CI 2-sided [-7.09 to 1.72]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -7.45, 95% CI 2-sided [-9.54 to -5.36]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -8.08, 95% CI 2-sided [-9.86 to -6.29]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -10.01, 95% CI 2-sided [-13.07 to -6.95]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -10.89, 95% CI 2-sided [-14.77 to -7.02]

24. Primary Outcome: Change From Baseline Over Time in CTx
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
pg/mL
  Change at Week 24: number analyzed (Participants) | 18
  Change at Week 24 | 343.38 (135.575)
  Change at Week 48 | 41.45 (61.062)
  Change at Week 72: number analyzed (Participants) | 19
  Change at Week 72 | -61.96 (63.458)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | -68.62 (63.152)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | -53.41 (50.545)
  Change at Week 144: number analyzed (Participants) | 19
  Change at Week 144 | -97.46 (55.670)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p = 0.0113, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 343.38, 95% CI 2-sided [77.66 to 609.11]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p = 0.4972, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 41.45, 95% CI 2-sided [-78.23 to 161.13]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p = 0.3288, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -61.96, 95% CI 2-sided [-186.34 to 62.41]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p = 0.2772, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -68.62, 95% CI 2-sided [-192.39 to 55.16]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p = 0.2907, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -53.41, 95% CI 2-sided [-152.47 to 45.66]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p = 0.0800, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = -97.46, 95% CI 2-sided [-206.57 to 11.65]

25. Primary Outcome: Change From Baseline Over Time in P1NP
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | KRN23
Number analyzed (Participants) | 20
ng/mL
  Change at Week 24 | 72.45 (16.962)
  Change at Week 48 | 44.40 (7.175)
  Change at Week 72 | 28.30 (7.684)
  Change at Week 96: number analyzed (Participants) | 19
  Change at Week 96 | 27.02 (6.739)
  Change at Week 120: number analyzed (Participants) | 19
  Change at Week 120 | 13.02 (8.359)
  Change at Week 144: number analyzed (Participants) | 19
  Change at Week 144 | 43.12 (33.717)
Statistical Analysis 1: Comparison: KRN23; Change at Week 24; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 72.45, 95% CI 2-sided [39.21 to 105.70]
Statistical Analysis 2: Comparison: KRN23; Change at Week 48; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 44.40, 95% CI 2-sided [30.34 to 58.47]
Statistical Analysis 3: Comparison: KRN23; Change at Week 72; Test type: Superiority; p = 0.0002, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 28.30, 95% CI 2-sided [13.24 to 43.37]
Statistical Analysis 4: Comparison: KRN23; Change at Week 96; Test type: Superiority; p < 0.0001, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 27.02, 95% CI 2-sided [13.81 to 40.22]
Statistical Analysis 5: Comparison: KRN23; Change at Week 120; Test type: Superiority; p = 0.1195, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 13.02, 95% CI 2-sided [-3.37 to 29.40]
Statistical Analysis 6: Comparison: KRN23; Change at Week 144; Test type: Superiority; p = 0.2009, GEE — [p-value comment as in outcome 10, analysis 2]; LS Mean = 43.12, 95% CI 2-sided [-22.96 to 109.20]

ADVERSE EVENTS:
Time Frame: Screening through the end of study plus 4-8 weeks. The mean duration of burosumab exposure was 165.6 weeks (range: 68-184 weeks).
Arm/Group | KRN23
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRN23 (N=20)
Hereditary Non-Polyposis Colorectal Cancer Syndrome (Congenital, familial and genetic disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
Medical Device Site Joint Infection (Infections and infestations) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemianaesthesia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRN23 (N=20)
Atrial Fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Vertigo Positional (Ear and labyrinth disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 2
Conjunctival Haemorrhage (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Visual Impairment (Eye disorders) | 1
Vitreous Floaters (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Faecal Incontinence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Intestinal Dilatation (Gastrointestinal disorders) | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1
Large Intestinal Stenosis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Pancreatic Calcification (Gastrointestinal disorders) | 1
Pancreatic Duct Dilatation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 1
Cyst (General disorders) | 1
Fatigue (General disorders) | 4
Gravitational Oedema (General disorders) | 1
Injection Site Erythema (General disorders) | 3
Injection Site Pain (General disorders) | 1
Injection Site Reaction (General disorders) | 4
Medical Device Site Pain (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Tenderness (General disorders) | 1
Ampulla Of Vater Stenosis (Hepatobiliary disorders) | 1
Biliary Dilatation (Hepatobiliary disorders) | 1
Hepatic Steatosis (Hepatobiliary disorders) | 2
Seasonal Allergy (Immune system disorders) | 2
Arthritis Infective (Infections and infestations) | 1
Breast Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 3
Gingivitis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Incision Site Infection (Infections and infestations) | 1
Infected Bite (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Lyme Disease (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 7
Otitis Externa (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Sinusitis Bacterial (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 2
Tooth Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 5
Urinary Tract Infection (Infections and infestations) | 2
Urinary Tract Infection Enterococcal (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 6
Femur Fracture (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 2
Procedural Hypertension (Injury, poisoning and procedural complications) | 1
Procedural Nausea (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 3
Tooth Injury (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Amylase Increased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Cholesterol Increased (Investigations) | 1
Blood Iron Decreased (Investigations) | 1
Blood Pressure Decreased (Investigations) | 1
Eosinophil Count Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 2
Haemoglobin Decreased (Investigations) | 1
Lipase Increased (Investigations) | 1
Oxygen Saturation Decreased (Investigations) | 1
Smear Cervix Abnormal (Investigations) | 1
Urine Electrophoresis Abnormal (Investigations) | 1
Weight Decreased (Investigations) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 1
Cervical Radiculopathy (Nervous system disorders) | 1
Cubital Tunnel Syndrome (Nervous system disorders) | 1
Disturbance In Attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Fine Motor Skill Dysfunction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 2
Nerve Compression (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Peroneal Nerve Palsy (Nervous system disorders) | 1
Restless Legs Syndrome (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Sinus Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Mental Status Changes (Psychiatric disorders) | 1
Bladder Prolapse (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hypercalciuria (Renal and urinary disorders) | 1
Nephrocalcinosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Renal Mass (Renal and urinary disorders) | 1
Urethral Stenosis (Renal and urinary disorders) | 1
Urinary Hesitation (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1
Menopausal Symptoms (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Scrotal Oedema (Reproductive system and breast disorders) | 1
Testicular Swelling (Reproductive system and breast disorders) | 1
Uterine Cervical Squamous Metaplasia (Reproductive system and breast disorders) | 1
Vaginal Prolapse (Reproductive system and breast disorders) | 1
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1
Vulvovaginal Pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Ophthalmic Fluid Drainage (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02312687/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT02312687/SAP_001.pdf